CLINICAL TRIAL: NCT04331093
Title: A Single-cencer,Phase II Study of Neoadjuvant SHR-1210 Plus Apatinib for Resectable Stage III-IV Acral Melanoma
Brief Title: Neoadjuvant SHR-1210 Plus Apatinib for Resectable Stage III-IV Acral Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Di Wu (Other)
Responsible Party: Sponsor-Investigator, Di Wu, professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k2020033
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Acral Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- resectable stage III-IV Acral melanoma (Experimental)
  Interventions: Drug: SHR-1210+Apatinib

INTERVENTIONS:
Drug: SHR-1210+Apatinib — Drug: SHR-1210 SHR-1210 will be administered as a 30-minute IV infusion Q2W at a dose of 200mg
  Drug: Apatinib Apatinib tablet will be administered orally,once daily until progression

SUMMARY:
Acral melanoma is a melanoma that affects acral areas of the skin, which is the most prevalent site of melanoma in non-Caucasians.Data in this subgroup is scarce.This study is to evalueate the efficiency and safety of Neoadjuvant SHR-1210 plus apatinib in this particular group,menawhile to determine the predictive value for efficiency of several biomarkers.

DETAILED DESCRIPTION:
SHR-1210 is a humanized monoclonal antibody against Programmed death 1(PD-1). Apatinib is a new kind of selective Vascular Endothelial Growth Factor Receptor 2(VEGFR-2) tyrosine kinase inhibitor (TKI).

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years. 2. Clinically diagnosed or pathologically diagnosed, resectable stage III-IV Acral melanoma with at least one measurable lesion that has not been treated locally (according to RECISTv1.1, this measurable lesion is spiral CT (Or MRI scan with a long diameter ≥10mm or an enlarged lymph node with a short diameter ≥15mm), patients with metastasis can also be enrolled; 3. Have not received any anti-tumor medication before. 4. ECOG score is 0 or 1. 5. Tumor tissue specimens must be provided for genetic testing (preoperative biopsy / intraoperative tissue removal).

6. Expected survival time ≥ 12 weeks. 7. The level of organ function must meet the following requirements (7 days before randomization):

* Peripheral blood: absolute neutrophil count (≥) 1.5 × 109 / L, platelet count (≥) 100 × 109 // L, hemoglobin (Hb) ≥9g / dL (no blood transfusion within 14 days before detection);

  * Liver: serum total bilirubin (≤) 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN (or AST, ALT ≤ 5 × ULN);

    * Serum creatinine ≤1.5 × ULN or endogenous creatinine clearance ≥50mL / min (using Cockcroft-Gault formula); ④. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (only applicable to patients who have not received anticoagulant therapy and received anticoagulant therapy, and anticoagulant drugs should meet the treatment requirements);

      ⑤. Cardiac function is normal, that is, the result of ECG is normal or has no clinical significance. Left ventricular ejection fraction (LVEF) of cardiac ultrasound examination is> 50%.

      8. Women of childbearing age must have a negative pregnancy test within 7 days before treatment; males of reproductive capacity or women who are at risk of pregnancy must use effective contraception throughout the study period and continue contraception for 3 months after the end of treatment.

      9. Can swallow pills normally. 10. Voluntarily participate in the research and sign the informed consent form, with good compliance and willingness to cooperate with the follow-up.

Exclusion Criteria:

1. Patients who have been treated with anti-PD-1, anti-PD-L1, VEGFRTKI;
2. Patients who are participating or are participating in clinical studies of other drugs or treatments, within 4 weeks before enrollment (prior to randomization);
3. Patients who received major surgery, vaccines, and systemic hormone therapy within 4 weeks before the study began; and patients who received radiation therapy within 2 weeks;
4. In the past 3 years, other malignancies other than acral or mucosal melanoma, except for cured skin basal cell carcinoma, skin squamous cell carcinoma, early prostate cancer and cervical cancer;
5. Receive hematopoietic stimulating factors (such as granulocyte colony stimulating factor (G-CSF) and erythropoietin) within 1 week before the start of the study.
6. HIV positive test;
7. Patients with active hepatitis B or C:

   ①. In the case of HBsAg or HBcAb positive, additional HBVDNA testing (results above the lower limit of detection specified by the study site).

   ②. In the case of HCV antibody positive, perform additional HCVRNA detection.
8. Urine routine indicates urinary protein ≥ ++ and it has been confirmed that the amount of urinary protein in 24 hours is> 1.0g;
9. Suffering from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
10. Pleural effusion or ascites with clinical symptoms and symptomatic treatment;
11. People with ocular shape and central nervous system (CNS) metastasis;
12. Have a history of active tuberculosis;
13. Have any uncontrollable clinical problems, including but not limited to:

    ①. Have autoimmune disease, or have a history of autoimmune disease or a syndrome requiring systemic treatment with steroids / immunosuppressants, such as pituitary inflammation, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism and thyroid Hypofunction

    ②. The following occurred within the first 6 months of randomization: 1) deep vein thrombosis or pulmonary embolism; 2) percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; 3) cerebrovascular accident, Transient ischemic attack.

    ③. Other serious and uncontrolled companion diseases that may affect the compliance of the agreement or the interpretation of the results, including active opportunistic or progressive (severe) infection, uncontrolled diabetes, cardiovascular disease (graded by the New York Heart Association) System-defined grade III or IV heart failure, grade II heart block, myocardial infarction in the past 6 months, unstable arrhythmia or unstable angina, cerebral infarction in the past three months, etc.). Or lung disease (history of interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm);
14. Patients with any condition that affects swallowing the drug, and any condition that affects the absorption of the research product in vivo, including any type of gastrointestinal resection or surgery;
15. Previous stem cell transplant or organ transplant;
16. Women with childbearing potential or pregnant or lactating women with a positive serum or urine pregnancy test within 7 days before the start of treatment;
17. Previously addicted to antipsychotic drugs, cannot be quit, or have a history of mental illness;
18. Other serious, acute or chronic medical conditions or laboratory abnormalities may increase the risks associated with participating in the research or may interfere with the interpretation of the research results by investigators;
19. Other conditions that the researchers consider to be non-compliant or not applicable to participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
pCR | 3 months
  Pathological complete response rate

SECONDARY OUTCOMES:
npCR | 3 months
  Near pathological complete response rate
ORR | 3 months
  Objective response rate
3 Year RFS | 3 years
  Recurrence free survival in 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China